CLINICAL TRIAL: NCT01062152
Title: Phase 1 Dose-Ranging Study of Ezatiostat Hydrochloride (Telintra®, TLK199 Tablets)in Combination With Lenalidomide (Revlimid®)in Patients With Non-Deletion(5q) Low to Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Dose-Ranging Study of Telintra® Tablets + Revlimid® in Patients With Non-Deletion (5q) Low to Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.1104
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Hematology; MDS; Myelodysplastic Syndrome; Low risk MDS; Patients with non-deletion(5q); Non-deletion 5q; Non del(5q); Revlimid; lenalidomide; Telintra; ezatiostat hydrochloride; ezatiostat; TLK199; Glutathione; Glutathione analog; Glutathione Transferase; Glutathione Transferase inhibitor; Glutathione Transferase P1-1 inhibitor; GSTp1-1 inhibitor; Apoptosis; Differentiation; Enzyme inhibitor
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Revlimid® in Combination with Telintra ® (Experimental): Lenalidomide (Revlimid®) followed by Telintra® until MDS progression or lack of efficacy.
  Interventions: Drug: Ezatiostat Hydrochloride; Drug: Lenalidomide (Revlimid®)

INTERVENTIONS:
Drug: Ezatiostat Hydrochloride — Starting dose 2000 mg orally in divided doses twice daily (1000 mg in AM & 1000 mg in PM) x 21 days with one week off therapy in a 4-week cycle.
Drug: Lenalidomide (Revlimid®) — 10 mg orally per day in one AM dose x 21 days with one week off therapy in a 4-week cycle.

SUMMARY:
This is an open label, multicenter Phase 1 dose escalation study evaluating five doses of ezatiostat in combination with lenalidomide in patients with non-del(5q) low to intermediate 1 risk MDS. The HI-E, HI-N, HI-P rates [by International Working Group (IWG) 2006 criteria] and safety of each treatment group will be evaluated to select the optimal dose of ezatiostat in combination with lenalidomide for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of primary or de novo MDS using WHO classification
* Non-del(5q) low or Intermediate-1risk MDS
* ECOG performance status of 0-1
* Documented significant cytopenia for at least 2 months
* Must have discontinued growth factors (EPO, G-CSF, GM-CSF) for at least 21 days prior to study entry
* All study participants must be registered into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist®
* Females of childbearing potential should have two negative serum pregnancy tests with a sensitivity of at least 50 mIU/mL. The first test should be performed within 10-14 days, and the second test within 24 hours of prescribing lenalidomide (prescriptions must be filled within seven days)

Exclusion Criteria:

* Known hypersensitivity to Telintra™ (intravenous or oral)
* Known prior therapy with or hypersensitivity to thalidomide or lenalidomide
* Prior allogenic bone marrow transplant for MDS
* History or prior malignancy

  * Except for treated carcinoma of uterine cervix, basal cell or squamous cell skin cancer, or other cancers (e.g. breast, prostate) for which patient has been disease-free for at least 3 years.
* MDS evolving from:

  * A pre-existing myeloproliferative disorder
  * An autoimmune disease
  * Secondary to prior treatment with radiation or chemotherapy
* History of MDS IPSS score>1.0
* Pregnant or lactating women
* Leptomeningeal or leukemic meningitis
* Prior treatment with DNA methyltransferase inhibitors (DMTI) [e.g., azacitadine, decitabine, etc.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of ezatiostat in combination with lenalidomide | 2 years
To determine the safety of ezatiostat in combination with lenalidomide | 2 years

SECONDARY OUTCOMES:
To determine the efficacy of ezatiosate in combination wiht lenalidomide in patients with non-del(5q) low to intermediate-1 risk of MDS | 2 years
Hematologic Improvement-Erythroid (HI-E) rate | 2 years
Hematologic Improvement-Neutrophil (HI-N) rate | 2 years
Hematologic Improvement-Platelet (HI-P) rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail Brown, M.D., Study Director — Telik
Locations (9):
- United States (9):
  - Mayo Clinic, Phoenix, Arizona
  - Loyola University Chicago Cardinal Benardin Cancer Center, Maywood, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - MDAnderson, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas

REFERENCES:
- [Derived] Raza A, Galili N, Mulford D, Smith SE, Brown GL, Steensma DP, Lyons RM, Boccia R, Sekeres MA, Garcia-Manero G, Mesa RA. Phase 1 dose-ranging study of ezatiostat hydrochloride in combination with lenalidomide in patients with non-deletion (5q) low to intermediate-1 risk myelodysplastic syndrome (MDS). J Hematol Oncol. 2012 Apr 30;5:18. doi: 10.1186/1756-8722-5-18. PMID 22546242